CLINICAL TRIAL: NCT00539656
Title: Transplantation of Expanded and Unexpanded Umbilical Cord Blood Units Following Myeloablative Chemotherapy for Hematologic Malignancies
Brief Title: Transplantation of Umbilical Cord Blood Following Chemotherapy for Blood Cancers
Acronym: Cord Blood
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The manufacturer discontinued necessary reagents.
Sponsor: Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins (Other)
Collaborators: Children's Cancer Foundation (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: J0606; NA_00001903 (Other: JHM IRB); M052663 (Other Grant/Funding Number: Children's Cancer Foundation)
Record Dates: First submitted 2007-10-02; First posted 2007-10-04 (Estimated); Results first posted 2019-04-03 (Actual); Last update posted 2020-02-18 (Actual); Status verified 2020-02

CONDITIONS: Acute Myeloid Leukemia; Leukemia, Lymphoblastic, Acute; Leukemia, Bilineage, Acute; Leukemia, Myeloid, Chronic
Keywords: Cord blood stem cell transplantation; Ex vivo expansion; Alternative donor
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Leukemia, Myelogenous, Chronic, BCR-ABL Positive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Receive two cord blood units (Experimental): One cord blood unit will be thawed on day -14 before transplantation and selected using the CliniMACS for primitive cells that express CD133. These cells will be expanded ex vivo for a total of 14 days, using a two-stage procedure. On Day 0 the expanded cells will be harvested, washed three times with CliniMACS buffer (Miltenyi) plus 1% HSA per standard laboratory and clinical practice and the expanded cell product will be infused to a patient who has been prepared with a standard, myeloablative preparative regimen. A second, unexpanded, cord blood product will be infused on Day +1 for safety.
  Interventions: Biological: Ex vivo expansion of cord blood

INTERVENTIONS:
Biological: Ex vivo expansion of cord blood — Day 0: the expanded cell product will be infused to patient; Day +1: A second, unexpanded, cord blood product will be infused
  Other Names: Miltenyi CliniMACS CD133

SUMMARY:
This study is to evaluate the safety of transplantation of two cord blood products, including toxicities in patients following high-dose, myeloablative chemotherapy for blood malignancies. It is also to determine if the use of two cord products results in an improvement in neutrophil engraftment.

DETAILED DESCRIPTION:
The success of BMT as a curative option for patients with malignancies is frequently limited by the inability to identify an appropriate donor in time for transplantation.

Transplantations utilizing umbilical cord blood stem cells are increasingly successful. Data suggest that there are fewer and less developed T-cells in cord products when compared to bone marrow and so are likely to produce less graft-vs.-host disease (GVHD) even in the mismatched setting. In addition, the grafts are easily available second to the ease of collection as compared with other sources such as bone marrow and peripheral blood stem cells (PBSCs). The ability to build cord blood repositories containing samples with HLA types from minorities has and will continue to increase the likelihood of finding suitable products for under represented minorities such as African-Americans, Hispanic populations and mixed ethnic populations.

Unfortunately, limitations remain, secondary to the time to engraftment when the cell dose is less than optimal, resulting in delayed or failed engraftment. In addition, increased cell dose appears to be associated with disease free survival. Therefore, this modality of transplant is generally limited to smaller patients. This protocol evaluates the infusion and engraftment of two cord blood products - one that has been expanded ex vivo and one that has not been expanded following myeloablative chemotherapy for the treatment of hematological malignancies.

Primary Objective:

-To evaluate the safety of transplantation of two cord products including an expanded unit including infusional toxicities and potential immunologic competition.

Secondary Objective:

-To determine if the use of two cord products results in an improvement in neutrophil engraftment (ANC>500) in subjects as demonstrated by engraftment <=21 days.

Tertiary Objectives:

Patients will be compared with patients participating in other trials at our institution and to those who receive therapy as per standard of care.

* To evaluate the rate, extent, and durability of hematopoietic reconstitution and in particular to determine the relative contribution of each cord unit in early engraftment and long-term engraftment
* To estimate the rate and severity of graft-vs-host disease
* To estimate the rates of infectious complications
* To obtain preliminary data regarding disease-free and overall survival
* To collect samples for future studies of immune reconstitution and for future studies in the laboratory regarding disease and the immune system

We will be able to track the fate of both the unmanipulated and expanded CB progenitors by evaluating differences in the cord products and the recipient by evaluation of sex mismatch, HLA type and/or restriction length polymorphisms (RFLPs). If the expanded CB cells are detected in the patients long-term, this will give us confidence to use expanded CB as the sole hematopoietic progenitor cell support, in future studies.

The major risk is non-engraftment of either one or both of the cord blood units. Non-engraftment of one of the units may lead to prolonged cytopenia and a marked increased risk for infection. Failure of either unit to engraft as defined as failure to detect cells from either cord blood product at Day +60 is likely to result in the death of the subject. There is the possibility of failure of long-term engraftment from both cords. This would be fatal unless an alternative donor option was identified or the unlikely event of autologous reconstitution of bone marrow. There is a possibility of an immune competition of both cord blood products . This could result in the loss of the cord product that would have been responsible for long term engraftment. There is a possibility of the expanded cord product to fail release testing. In this event, only the unexpanded cord would be infused and would likely result in delayed engraftment.

As with all cellular products there are risks associated with the infusion including but not limited to anaphylaxis, transfusion reaction, hemolysis, side-effects of the DMSO that the product is stored in (bradycardia, hypothermia, neurologic changes). The expanded product will be washed however there remains a small chance that a small amount of growth factor remains. The risk associated with these will be allergic.

Busulfan toxicity

1. Nausea and vomiting
2. Myeloablation
3. Pulmonary complications
4. Seizures
5. Other toxic effects which may be produced by Busulfan erythematous skin rash, hyperpigmentation, hepatic dysfunction, amenorrhea, testicular atrophy, gynecomastia, myasthenia symptoms, cataract and atrophic bronchitis associated with cytologic dysplasia.

Cyclophosphamide Toxicity

1. Leukopenia, anemia
2. Alopecia
3. Nausea, vomiting, increased AST, ALT, mucositis, diarrhea
4. Headache, dizziness
5. Cardiac necrosis rarely with high dose cyclophosphamide
6. Hemorrhagic cystitis, SIADH
7. Teratogenic, may cause secondary neoplasms, anaphylaxis (rare)
8. Fluid retention.
9. Cardiomyopathy.
10. Hemorrhagic Cystitis.

At the doses used for uroprotection mesna is virtually non-toxic. However, adverse effects which may be attributable to mesna include nausea and vomiting, diarrhea, abdominal pain, altered taste, rash, urticaria, headache, joint or limb pain, hypotension and fatigue.

Total Body Irradiation Toxicity:

1. Nausea and Vomiting
2. Alopecia
3. Parotitis and Pancreatitis
4. Diarrhea
5. Fever
6. Erythema
7. Hyperpigmentation
8. Mucositis
9. Late Effects - cataract formation, growth retardation, carcinogenesis and the probability of sterilization.

ELIGIBILITY:
Inclusion Criteria:

* Patient must have two cord units available. Units must be minimally matched to the subject at 4/6 antigens (HLA Class I (A or B) and Class II (DRB1) - units must have at lease one HLA DRB1 matched allele) and at least one unit must contain a minimum of 1.0 x 107 Total Nucleated Cells /Kg but neither unit may have > 5 x 107Total Nucleated Cells /Kg. (The feasibility of using particular units will be discussed with the Principal Investigators)
* Disease status precludes waiting to identify a suitably HLA matched unrelated donor
* Patients must have a diagnosis of one of the following:

  * AML
  * refractory AML
  * Secondary AML
  * ALL in CR2 with high-risk features such as short CR1 and/or high-risk cytogenetics
  * ALL in CR1 following initial induction failure
  * Acute mixed lineage leukemia
  * CML beyond chronic phase 1.
  * Lymphoma (Hodgkins or Non-Hodgkins) ineligible for Autologous-BMT
  * Myelodysplastic Syndrome
* Able to provide informed consent or parent/guardian able to provide informed consent.

Exclusion Criteria:

* Consenting 5/6 or 6/6 HLA matched related donor available
* Single cord blood product with cell count >5 x10E7 Total Nucleated Cells/kg
* Poor Performance Status: ECOG performance status >= 2 (Karnofsky or Lansky Play performance<70).
* Poor Cardiac Function (obtained within 3 weeks of the start of transplant): Left ventricular ejection fraction <= 45% as determined by MUGA or ECHO. For pediatric patients LVEF < 45 % or a Shortening Fraction below normal limits for age.
* Poor Pulmonary Function (obtained within 3 weeks of the start of transplant):

  * FEV1 and FVC <50% of predicted for patients who have not received thoracic or mantle irradiation.
  * For patients who have received thoracic or mantle irradiation, FEV1 and FVC <= 75% of predicted or DLCO <= 50% of predicted
  * For children unable to perform PFTs second to developmental stage, Pulse oximetry <= 85% on RA
* Poor Liver Function (obtained within 1 week of the start of transplant): Bilirubin >= 2.0 mg/dl. (with the exception of patients whose hyperbilirubinemia is the result of Gilbert's disease)
* Poor Renal Function (obtained within 3 weeks of the start of transplant): Corrected CrCl < 60 mg/min. CrCl will be estimated by the Schwartz formula. A measured CrCl or a GFR may be substituted to determine the subject's CrCl
* HIV Infection: Patients who are HIV positive. (The role of allogenic transplant in HIV+ individuals has not been studied)
* Pregnancy: Patients who are pregnant. (The chemotherapeutic agents used in bone marrow transplant are teratogenic)
* Uncontrolled viral, bacterial or fungal infections
* Patients with symptoms consistent with RSV, influenza A, B or parainfluenza at the time of enrollment on this study will be assayed for the above viruses and if positive are not eligible for the trial until are no longer symptomatic (patients may have continued assay positivity for a period of time post resolution of symptoms second to the nature of the assay)
* Presence of concomitant medication or incident condition that would create an unreasonable risk for the subject to participate in this study as determined by the investigators (Primary or co-investigators).
* Patients with known intolerance to or contraindication for any agent that will be used in the subject's proposed myeloablative or required supportive care regimen.

Ages: 6 Months to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2007-12-20 (Actual); Primary Completion 2009-10-20 (Actual); Study Completion 2009-10-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allen R. Chen, MD,PhD. MHS, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins Hospital, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Single Arm: Patients with a hematologic malignancy who are candidates for myeloablative allogeneic BMT but lack an available matched sibling or unrelated marrow donor are eligible for this study if they have two suitably matched cord blood products with an adequate (1 x 10e7 TNC/kg IBW) but suboptimal (<5 x 10e7 TNC/kg IBW) cell dose. Eligible diagnoses include AML, MDS, ALL after failure of at least one regimen, mixed lineage leukemia, CML beyond first chronic phase, and lymphoma ineligible for autologous transplantation.
Period: Overall Study
Arm/Group | Single Arm
Started | 3
Completed | 3
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: Patients with a hematologic malignancy who are candidates for myeloablative allogeneic BMT but lack an available matched sibling or unrelated marrow donor are eligible for this study if they have two suitably matched cord blood products with an adequate (1 x 10e7 TNC/kg IBW) but suboptimal (<5 x 10e7 TNC/kg IBW) cell dose.
  One cord blood unit is expanded beginning 14 days before graft infusion (6 or 7 days before the start of the preparative regimen). Patients receive a standard myeloablative preparative regimen. The expanded cord blood unit is infused on day 0 and the unmanipulated cord blood unit is expanded on day 1.
Arm/Group | Single Arm
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 0
Age, Continuous [Median (Full Range); unit: years] | 37 [18 to 38]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Toxicities Related to Infusion of Expanded Cord Blood Products
Time Frame: 7 days
Measure: Count of Participants; unit: Participants
Arm/Group | Receive Two Cord Blood Units
Number analyzed (Participants) | 3
Participants | 0

2. Primary Outcome: Neutrophil Engraftment Within 21 Days
Description: Number of participants who reached 3 consecutive days with ANC > 500
Time Frame: 21 days
Measure: Count of Participants; unit: Participants
Arm/Group | Receive Two Cord Blood Units
Number analyzed (Participants) | 3
Participants
  Engrafted by day 21 | 1
  Not engrafted by day 21 | 2

3. Secondary Outcome: Non-relapse Mortality
Description: Number of participants who died without relapse in less than 100 days.
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Receive Two Cord Blood Units
Number analyzed (Participants) | 3
Participants | 1

ADVERSE EVENTS:
Time Frame: up to 100 days
Description: Neutrophil count was followed based on regular lab assessments
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 1/3
Serious Adverse Events (participants affected / at risk) | 1/3
Other Adverse Events (participants affected / at risk) | 3/3
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Single Arm (N=3)
ARDS (Respiratory, thoracic and mediastinal disorders) | 1 (1) — Death due to ARDS, grade 5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=3)
Neutropenia (Blood and lymphatic system disorders) | 3 — low neutrophils

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes